CLINICAL TRIAL: NCT02211417
Title: A Randomised, Double-Blind, Placebo-Controlled, Phase II Study to Assess the Efficacy and Safety of Orally Administered DS107G to Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Oral DS107 in Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dignity Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS107G-02
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 8,11,14-Eicosatrienoic Acid; Gelatin; Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral DS107 2g (Experimental): Oral DS1072g, 4 x 500mg capsules administered orally once a day
  Interventions: Drug: Oral DS107
- Placebo (Placebo Comparator): Placebo capsules matching Oral DS107 capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral DS107
  Other Names: DGLA (Dihomo-gamma-linolenic acid) 500 mg gelatin capsule
  Arms: Oral DS107 2g
Drug: Placebo
  Other Names: Liquid paraffin capsule to mimic Oral DS107 500 mg gelatin capsule
  Arms: Placebo

SUMMARY:
This study will compare the safety and efficacy of Oral DS107 (2 g) to placebo in patients with moderate to severe atopic dermatitis.

Oral DS107 (2 g) will be orally administered for 8 weeks, and will be compared against placebo.

This study will enroll approximately 100 adult patients.

DETAILED DESCRIPTION:
Subjects will come to the clinic on 6 occasions: at screening, baseline, week 2, week 4, week 8 (end of treatment/early termination) and week 10 (follow-up). The primary efficacy variable will be the IGA. Secondary efficacy variables will include IGA (Investigator's Global Assessment), SCORAD (Scoring Atopic Dermatitis) Visual Analog Scale (VAS), EASI, BSA (Body Surface Area), POEM (Patient Orientated Eczema Measure), DLQI (Dermatology Life Quality Index).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 years and older.
* Moderate to severe atopic dermatitis.

Exclusion Criteria:

* Clinically significant impairment of renal or hepatic function.
* History of hypersensitivity to any substance in Oral DS107 or placebo capsules.
* Treatment with any experimental drug within 30 days prior to Day 0 visit (baseline).
* Excessive sun exposure, use of tanning booths or other ultraviolet (UV) light sources and/or is planning a trip to sunny climate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Climax, Ph.D., Study Chair — Dignity Sciences Ltd.
Locations (14):
- United States (8):
  - Dignity Sciences investigational site, Arlington Heights, Illinois
  - Dignity Sciences investigational site, West Dundee, Illinois
  - Dignity Sciences investigational site, Warren, Michigan
  - Dignity Sciences investigational site, Verona, New Jersey
  - Dignity Sciences investigational site, New York, New York
  - Dignity Sciences investigational site, Rochester, New York
  - Dignity Sciences investigational site, Hazleton, Pennsylvania
  - Dignity Sciences investigational site, Philadelphia, Pennsylvania
- Canada (6):
  - Dignity Sciences investigational site, Calgary, Alberta
  - Dignity Sciences investigational site, Edmonton, Alberta
  - Dignity Sciences investigational site, Markham, Ontario
  - Dignity Sciences investigational site, Windsor, Ontario
  - Dignity Sciences investigational site, Drummondville, Quebec
  - Dignity Sciences investigational site, Montreal, Quebec

REFERENCES:
- [Background] Scollan ND, Choi NJ, Kurt E, Fisher AV, Enser M, Wood JD. Manipulating the fatty acid composition of muscle and adipose tissue in beef cattle. Br J Nutr. 2001 Jan;85(1):115-24. doi: 10.1079/bjn2000223. PMID 11227040
- [Background] Kawashima H, Toyoda-Ono Y, Suwa Y, Kiso Y. Subchronic (13-week) oral toxicity study of dihomo-gamma-linolenic acid (DGLA) oil in rats. Food Chem Toxicol. 2009 Jun;47(6):1280-6. doi: 10.1016/j.fct.2009.03.001. Epub 2009 Mar 9. PMID 19275928
- [Background] Makrides M, Simmer K, Neumann M, Gibson R. Changes in the polyunsaturated fatty acids of breast milk from mothers of full-term infants over 30 wk of lactation. Am J Clin Nutr. 1995 Jun;61(6):1231-3. doi: 10.1093/ajcn/61.6.1231. PMID 7762522
- [Background] Teraoka N, Kawashima H, Shiraishi-Tateishi A, Tanaka T, Nakamura J, Kakutani S, Kiso Y. Oral supplementation with dihomo-gamma-linolenic acid-enriched oil altered serum fatty acids in healthy men. Biosci Biotechnol Biochem. 2009 Jun;73(6):1453-5. doi: 10.1271/bbb.90112. Epub 2009 Jun 7. PMID 19502748
- [Background] Tanaka T, Kakutani S, Horikawa C, Kawashima H, Kiso Y. Oral supplementation with dihomo-gamma-linolenic acid (DGLA)-enriched oil increases serum DGLA content in healthy adults. Lipids. 2012 Jun;47(6):643-6. doi: 10.1007/s11745-012-3664-3. Epub 2012 Mar 14. PMID 22411689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 countries at 17 sites.
Pre-assignment Details: A total of 102 patients were randomised. Patients were randomised (1:1) at baseline visit to either receive Oral DS107 capsules (2 g) or Placebo once daily for 8 weeks in a fasting state (minimum 8 hour fast).
Period: Overall Study
Arm/Group | Placebo | Oral DS107 2g
Started | 51 | 51
Completed | 36 | 35
Not Completed | 15 | 16
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population - The safety population was defined as all randomised patients who received at least one dose of the medication. Analysis was done according to the actual treatment patients received.
Groups:
- Oral DS107 2g: Oral DS107 2g, 4 x 500mg capsules administered orally once a day
- Total: Total of all reporting groups
Arm/Group | Placebo | Oral DS107 2g | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (15.7) | 35.7 (13.6) | 39.8 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 28 | 21 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 16 | 35
  White | 26 | 30 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving an Investigator's Global Assessment (IGA) of 0 (Clear) or 1 (Almost Clear) and a Decrease of at Least 2 Points in IGA at Week 8.
Description: The IGA is a global assessment of the current state of the disease. It is a 6-point morphological assessment of overall disease severity and will be determined according to the following definitions: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), 4 (severe) and 5 (very severe). The scale uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment. A decrease in IGA indicates a positive outcome for the participant.
Time Frame: Week 8
Population: ITT Population - The Intent-to-treat (ITT) population consisted of all randomised patients. Analysis was done according to the randomised treatment. This population was used for all efficacy analyses.
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
Proportion of participants | 0.12 | 0.22
Statistical Analysis 1: Comparison: Placebo vs Oral DS107 2g; Test type: Superiority; p = 0.057, Cochran-Mantel-Haenszel

2. Secondary Outcome: Change From Baseline in IGA at Week 2, 4 and 8.
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
units on a scale
  Week 2 | -0.2 (0.4) | -0.4 (0.7)
  Week 4 | -0.4 (0.6) | -0.9 (0.7)
  Week 8 | -0.9 (0.8) | -1.3 (1.2)

3. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) at Week 2, 4 and 8.
Description: EASI quantifies the severity of a patient's AD based on both lesion severity and the percent of BSA affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The severity of each sign is assessed using a 4-point scale (half points are permitted):
  * 0 = no symptoms
  * 1 = slight
  * 2 = moderate
  * 3 = marked
  A decrease in EASI score indicates a positive outcome for the participant.
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DS107G: Oral DS107 2g, 4 x 500mg capsules administered orally once a day
Arm/Group | Placebo | DS107G
Number analyzed (Participants) | 51 | 51
units on a scale
  Week 2 | -1.2 (3.6) | -2.8 (5.1)
  Week 4 | -5.2 (7.9) | -7.2 (8.5)
  Week 8 | -8.4 (9.5) | -9.4 (11.11)

4. Secondary Outcome: Proportion of Patients Achieving at Least a 1-point Decrease in IGA at Week 8.
Description: as for outcome 1
Time Frame: Up to 8 weeks.
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
Proportion of participants | 0.43 | 0.51

5. Secondary Outcome: Change From Baseline in the Patient Orientated Eczema Measure (POEM) at Week 2, 4 and 8.
Description: The Patient-Oriented Eczema Measure (POEM) is a self-assessment of disease severity by the patient. POEM has a maximum value of twenty-eight based on the patient's response to seven questions scored according to the following scale:
  * No Days = 0
  * 1-2 Days = 1
  * 3-4 Days = 2
  * 5-6 Days = 3
  * Everyday = 4
  POEM scale ranges from 0 to 28. 0 to 2 = clear or almost clear. 3 to 7 = mild eczema. 8 to 16 = moderate eczema. 17 to 24 = severe eczema. 25 to 28 = very severe eczema.
  Lower scores on the scale represent a better outcome for the patient.
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
score on a scale
  Week 2 | -3.5 (5.6) | -5.0 (5.6)
  Week 4 | -4.0 (6.5) | -6.9 (6.3)
  Week 8 | -5.0 (7.7) | -5.7 (6.5)

6. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Score at Week 2, 4 and 8.
Description: The DLQI is a simple 10-question validated questionnaire measuring the impact of a patients skin problem over a 1 week period, which was completed at each visit, except screening. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
score on a scale
  Week 2 | -3.6 (5.5) | -4.2 (5.5)
  Week 4 | -5.0 (6.0) | -6.5 (5.9)
  Week 8 | -4.9 (5.5) | -5.5 (7.0)

7. Secondary Outcome: Change From Baseline in Scoring of Atopic Dermatitis (SCORAD) at Week 2, 4 and 8.
Description: The SCORAD grading system was developed by the European Task Force on Atopic Dermatitis and has been a standard tool to assess the AD severity in clinical studies. Six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) was selected to evaluate the AD severity. The intensity of each item is graded using a 4-point scale:
  * 0 = No symptoms
  * 1 = Mild
  * 2 = Moderate
  * 3 = Severe The overall BSA affected by AD was evaluated (from 0 to 100%) and included in the SCORAD scores. Loss of sleep and pruritus were evaluated by patients on a visual analog scale (0-10). The sum of these measures represents the SCORAD which can vary from 0 to 103. A decrease in SCORAD indicates a positive outcome for the participant.
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
score on a scale
  Week 2 | -5.3 (8.7) | -6.6 (10.3)
  Week 4 | -10.6 (14.7) | -16.7 (15.5)
  Week 8 | -18.3 (18.4) | -21.1 (21.7)

8. Secondary Outcome: Change From Baseline in the Patient's Visual Analog Scale (VAS) Pruritus Score at Week 2, 4 and 8.
Description: The pruritus severity score was recorded with the SCORAD measurement and was evaluated as a separate endpoint. This was evaluated by asking subjects to indicate on the 10-cm scale (0-10) of the assessment form the point corresponding to the average value for the last three days/nights. A lower score represents a better outcome for the patient.
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
score on a scale
  Week 2 | -0.9 (2.1) | -1.6 (2.5)
  Week 4 | -1.1 (2.7) | -2.8 (2.9)
  Week 8 | -2.2 (3.3) | -2.8 (3.0)

9. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) at Week 2, 4 and 8.
Description: One patient's palm represents 1% of his/her total BSA. For all study visits except at screening, the BSA of involved skin will be measured with the SCORAD measurement and evaluated as a separate endpoint.
Time Frame: Baseline, Week 2, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
percentage of BSA
  Week 2 | -0.9 (4.9) | -1.3 (4.4)
  Week 4 | -3.6 (7.1) | -5.2 (7.3)
  Week 8 | -7.0 (9.6) | -9.6 (13.8)

10. Secondary Outcome: Number of Participants With TEAEs in Each Treatment Group
Description: Number of participants with at least 1 TEAE.
Time Frame: Up to 14 weeks
Population: The safety population was defined as all randomised patients who received at least one dose of the medication. Analysis was done according to the actual treatment patients received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral DS107 2g
Number analyzed (Participants) | 51 | 51
Participants | 24 | 37

ADVERSE EVENTS:
Time Frame: Up to 14 weeks.
Description: An adverse event was defined as any untoward medical occurrence in a patient administered a pharmaceutical product, without regard to the possibility of a causal relationship with this treatment.
Arm/Group | Placebo | Oral DS107 2g
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/51
Other Adverse Events (participants affected / at risk) | 23/51 | 37/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Oral DS107 2g (N=51)
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Oral DS107 2g (N=51)
Diarrhoea (Gastrointestinal disorders) | 4 | 16
Nausea (Gastrointestinal disorders) | 1 | 16
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 8
Vomiting (Gastrointestinal disorders) | 1 | 5
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 2
Anal Pruritus (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Faeces Soft (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4
Abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Skin Bacterial Infections (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated Partial Thromboplastin Time Abnormal (Investigations) | 0 | 1
Blood Test Abnormal (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Restless Leg Syndrome (Nervous system disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Premenstrual Cramps (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT02211417/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT02211417/SAP_001.pdf